CLINICAL TRIAL: NCT07096414
Title: Effect of Vitamin D3 Supplementation on Brain Waves in Male Epileptic Patients With Hypovitaminosis D: A Quantitative Electroencephalogram Analysis
Brief Title: Effect of Vitamin D3 Supplementation on Brain Waves in Male Epileptic Patients With Hypovitaminosis D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Sumayya Binte Abdur Razzaque, MD resident, Bangladesh Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5587
Record Dates: First submitted 2025-07-10; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy; Hypovitaminosis D
Keywords: Epilepsy; Vitamin D3; Hypovitaminosis D; QEEG; Brainwaves
MeSH Terms: conditions — Epilepsy; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Experimental study (Interventional, self-controlled trial) where 15 participants will be enrolled to compare their baseline data with post interventional data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Male epileptic patients with hypovitaminosis D (Experimental): 15 male epileptic patients with hypovitaminosis D will be supplemented with vitamin D orally 50,000 IU/week for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Administration of vitamin D3 capsule 50,000 IU/week for 8 weeks

SUMMARY:
This is an experimental study (interventional self-controlled trial, pretest-post test design). The goal of this clinical trial is to evaluate the effect of vitamin D3 supplementation on quantitative EEG in male epileptic patients with hypovitaminosis D.

. The main question it aims to answer is:

Vitamin D3 supplementation has effect on brain waves in male epileptic patients with hypovitaminosis D.

Researcher will compare the effect of Vitamin D3 supplementation on brain waves in male epileptic patients with hypovitaminosis D with their pre-intervention (baseline) condition on brain waves to assess whether there will be any improvement of brain electrical activity by quantitative electroencephalogram (QEEG).

Participants will:

Take Vitamin D3 orally for 8 weeks (50,000IU/week) Visit the medical university after 8 weeks for evaluation of serum 25 (OH) D level and quantitative electroencephalogram (QEEG) Must bring the empty strips of Vitamin D supplement with them during their visit

DETAILED DESCRIPTION:
This experimental study (self-controlled trial) will be conducted by the Department of Physiology, Bangladesh Medical University, Shahbag, Dhaka from March 2025-February 2026. For this study, a total number of 15 male patients with Epilepsy (age 20-40 years) will be enrolled as study participants according to selection criteria (Diagnosed male patients with Epilepsy by neurologist from the Out Patient Department of Department of Neurology by taking proper history of at least two unprovoked (or reflex) seizures occurring > 24 hours apart, from patients and eye witnesses, having Hypovitaminosis D (<30 ng/ml), Age: 20-40 years, BMI : 20 - 24 kg/m², On antiepileptic medication for 6 months to 2 years (enzyme inducing AEDs, e.g. Carbamazepine, Phenytoin, Phenobarbital), Without any medication that affect central nervous system other than antiepileptic drugs (Antidepressants, Antipsychotic, Anxiolytic, Anesthetic drugs), Apparently normal physical health ) At first baseline serum 25(OH) D level will be measured & baseline QEEG will be recorded. After that the participants will be supplemented vitamin D3 orally (50,000IU/week) for 8 weeks. After completion of 8 weeks, serum 25(OH) D level will be measured again & QEEG will be recorded.

To analyze brain electrical activities, the band power of alpha, beta, theta, and Delta brainwaves will be measured using an EEG Data gathering Device, the EEG Traveler BrainTech 32+ CMEEG-01 from India. The BT40 analysis software will be used to perform power spectral analysis of the EEG data. Mean ± SD will be used to express the data.

For statistical analysis, to compare the mean values between the pre intervention and post intervention sessions, paired t test will be done.The P value of ≤0.05 will be accepted as statistically significant. SPSS for Windows (version 25) will be used for the statistical analysis.

The findings of this study are expected to provide quantitative evidence regarding the neurophysiological effects of vitamin D3 supplementation in male epileptic patients with hypovitaminosis D.Also it could help people with epilepsy to lead healthier, more productive lives.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed male patients with Epilepsy by neurologist from the Out Patient Department of Department of Neurology, BMU by taking proper history of at least two unprovoked (or reflex) seizures occurring > 24 hours apart, from patients and eye witnesses.
* Hypovitaminosis D (<30 ng/ml)
* BMI : 20 - 24 kg/m²
* On antiepileptic medication for 6 months to 2 years (enzyme inducing AEDs, e.g. Carbamazepine, Phenytoin, Phenobarbital)
* Without any medication that affect central nervous system other than antiepileptic drugs (Antidepressants, Antipsychotic, Anxiolytic, Anesthetic drugs)
* Apparently normal physical health

Exclusion Criteria:

* Patients suffering from absence seizure
* Certain AEDs (Sodium valproate, Ethosuximide, Oxcarbazepine, Topiramate, Lamotrigine, Levetiracetam)
* Smoker
* Alcoholic
* Known hypersensitivity to vitamin D3
* Patients with hypertension
* Patient with Thyroid disorder
* Patient with Diabetes mellitus
* Patient with Renal Disease
* Patient with liver Disease
* Patient with hypercalcemia

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Vitamin D3 supplementation has positive effect on brain waves in male epileptic patients with hypovitaminosis D that can be proved by quantitative electroencephalogram. | 8 weeks
  15 male epileptic patients with serum 25(OH)D level less than normal, will be supplemented with vitamin D capsule 50,000 IU/WEEK for 8 weeks. That may have an effect on brain electrical activity (altering the power of different frequency brain waves) and ultimately change seizure frequency which can be assessed by quantitative EEG using Fast Fourier Transform method.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Sumayya Binte Abdur Razzaque, MBBS, MD Resident (Phase B), Principal Investigator — BMU
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No